CLINICAL TRIAL: NCT01690299
Title: A Phase 3B, Multicenter, Randomized, Placebo-Controlled, Double-Blind, Double-Dummy, Study Of The Efficacy And Safety Of Apremilast (CC-10004), Etanercept, And Placebo, In Subjects With Moderate To Severe Plaque Psoriasis
Brief Title: Phase 3b Safety and Efficacy Study of Apremilast to Treat Moderate to Severe Plaque-plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-010; 2012-000859-14 (EudraCT Number)
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis; Psoriatic Arthritis
Keywords: Psoriasis; arthritis; psoriatic; palmoplantar; scalp; psoriasis pill; psoriasis tablet; plaque psoriasis; plaque type psoriasis; moderate to severe plaque type psoriasis; psoriatic arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Arthritis | interventions — apremilast; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Apremilast 30 mg plus placebo injection (Experimental): Apremilast 30 mg tablets orally twice a day (BID) plus once weekly (QW) evaluator/subject-blinded subcutaneous (SC) saline (placebo) injections
  Interventions: Drug: Apremilast; Drug: Placebo injection
- Etanercept 50 mg plus placebo tablet (Experimental): Etanercept 50 mg evaluator/subject-blinded SC QW injections plus placebo tablets orally BID
  Interventions: Drug: Etanercept; Drug: Placebo tablet
- Oral placebo tablets plus SC placebo injections (Placebo Comparator): Identically matching placebo tablets and evaluator/subject-blinded SC injections
  Interventions: Drug: Placebo tablet; Drug: Placebo injection

INTERVENTIONS:
Drug: Apremilast — Apremilast 30 mg tablet orally BID
  Other Names: CC-10004; Otezla
  Arms: Apremilast 30 mg plus placebo injection
Drug: Etanercept — Etanercept 50 mg evaluator/subject-blinded SC QW injection
  Other Names: Enbrel
  Arms: Etanercept 50 mg plus placebo tablet
Drug: Placebo tablet — Placebo tablets BID
  Arms: Etanercept 50 mg plus placebo tablet; Oral placebo tablets plus SC placebo injections
Drug: Placebo injection — Once weekly evaluator/subject-blinded SC placebo (1 mL x 2 injections SC)
  Arms: Apremilast 30 mg plus placebo injection; Oral placebo tablets plus SC placebo injections

SUMMARY:
This study will test the clinical effectiveness and safety of apremilast compared with placebo as well as etanercept compared with placebo in the same group of patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a phase 3b, multicenter, randomized, placebo-controlled, double-blind, double-dummy, study of the efficacy and safety of apremilast, etanercept, and placebo, in adults with moderate to severe plaque psoriasis.

250 participants will be randomized 1:1:1 to the three treatment groups. All subjects will receive both tablets and injections through Week 16.

The study will consist of four phases:

* Screening Phase - up to 35 days
* Double-blind Placebo-controlled Phase - Weeks 0-16
* Apremilast Extension Phase - Weeks 16-104
* Post-treatment Observational Follow-up Phase

During the double-blind, placebo-controlled phase, subjects will receive treatment with one of the following:

* apremilast (APR) 30 mg tablets orally twice a day (BID) plus once weekly (QW) evaluator/subject-blinded subcutaneous (SC) saline (placebo) injections (1 mL x 2 injections SC), or
* etanercept (ETN) 50 mg evaluator/subject-blinded subcutaneous (SC) once weekly (QW) injections (2 x 25 mg) plus placebo tablets orally twice a day (BID), or
* placebo tablets and evaluator/subject-blinded subcutaneous (SC) saline (placebo) injections.

All subjects will be asked to participate in a 4-week Post-treatment Observational Follow-up Phase either upon completion of the study or upon discontinuation of investigational product for those subjects who terminate the study early.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ≥ 18 years of age
* Diagnosis of chronic, moderate to severe plaque psoriasis for at least 12 months prior to Screening, and a candidate for phototherapy and/or systemic (including etanercept) therapy
* Had an inadequate response, intolerance, or contraindication to at least 1 conventional systemic agent for the treatment of psoriasis.
* No prior exposure to biologics for treatment of psoriatic arthritis or psoriasis

Exclusion Criteria:

* Other than psoriasis, history of any clinically significant and uncontrolled systemic diseases; any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
* Pregnant or breast feeding.
* Have failed more than 3 systemic agents for treatment of psoriasis.
* History of allergy to any component of the investigational product (IP), including human immunoglobulin (Ig) proteins or allergy to etanercept.
* Hepatitis B surface antigen or anti-hepatitis C antibody positive at Screening.
* Latent, active tuberculosis (TB) or inadequately treated TB; nontuberculous mycobacterial infection or opportunistic infection (eg, cytomegalovirus, Pneumocystis carinii, aspergillosis, Clostridium difficile).
* Have a history of, or ongoing, chronic or recurrent infectious disease
* Have received, or are expected to receive, any live virus or bacterial vaccination within 3 months before first administration of IP, or through Week 20 during the study.
* Had a Bacillus Calmette-Guérin (BCG) vaccination within 1 year prior to screening.
* History of positive human immunodeficiency virus (HIV), or have congenital or acquired immunodeficiency (eg, common variable immunodeficiency disease).
* Active substance abuse or a history of substance abuse within 6 months prior to Screening.
* Malignancy or history of malignancy, except for treated [ie, cured] basal cell or squamous cell in situ skin carcinomas and cervical intraepithelial neoplasia [CIN] or carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years.
* Psoriasis flare or rebound within 4 weeks prior to Screening.
* Topical therapy within 2 weeks of randomization or systemic therapy for psoriasis within 4 weeks prior to randomization
* Use of phototherapy within 4 weeks prior to randomization or prolonged sun exposure or use of tanning booths or other ultraviolet (UV) light sources.
* Any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer).
* Prior treatment with apremilast or etanercept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2014-07-03 (Actual); Study Completion 2016-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (82):
- United States (31):
  - Arizona Research Center, Phoenix, Arizona
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - University of California Irvine-Department of Dermatology, Irvine, California
  - University of California San Diego Medical Center, San Diego, California
  - Horizons Clinical Research, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Florida Center for Dermatology, PA, Jacksonville, Florida
  - Florida Academic Dermatology Center, Miami, Florida
  - International Dermatology Research, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Atlanta Dermatology, Vein and Research Center, PC, Alpharetta, Georgia
  - NorthShore University HealthSystem, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dermatology and Advanced Aesthetics, Lake Charles, Louisiana
  - Lawrence Green, MD, LLC, Rockville, Maryland
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Robert Wood Johnson Medical School, Somerset, New Jersey
  - Forest Hills Dermatology Group, Forest Hills, New York
  - NYU Department of Dermatology, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennesse Clinical Research Center, Nashville, Tennessee
  - Teckton Research, Austin, Texas
  - The Education and Research Foundation, Lynchburg, Virginia
  - Virginia Clinical Research Inc, Norfolk, Virginia
  - Dermatology Associates of Seattle, Seattle, Washington
- Australia (6):
  - The Skin Centre, Benowa, Queensland
  - Sinclair Dermatology, East Melbourne, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
  - Gairdner Hospital, Victoria Park
  - Rheumatology unit Ward 5C Queen Elizabeth Hospital, Woodville
  - Veracity Clinical Research, Woolloongabba
- Belgium (3):
  - Cliniques Universitaires St-Luc, Brussels
  - University Hospital Ghent, Ghent
  - University Hospital of Liege CHU Liege, Liège
- Canada (5):
  - Eastern Canada Cutaneous Research Associates Ltd, Halifax, Nova Scotia
  - Skin Center for Dermatology, Peterborough, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - Siena Medical Research, Montreal, Quebec
  - Q & T Research Sherbrooke Inc., Sherbrooke, Quebec
- Czechia (6):
  - Dorothea, Kožní a korektivne dermatologické pracovište, Chomutov
  - Dermamedica, Náchod
  - Východoceské dermatologické centrum Homea s.r.o., Pardubice
  - Krajská nemocnice Pardubice, Kožní oddelení, Pardubice
  - Dermatovenerologicka ambulance, Svitavy
  - Koznia zilni ambulance, Ústí nad Labem
- Estonia (2):
  - South Estonian Hospital Ltd, Meegomäe Village, Võru County
  - Dermatology Clinic of Tartu University Hospital, Tartu
- Germany (14):
  - Psoriasis Study Center, Berlin
  - Dermatologische Praxis, Berlin
  - Klinische Forschung Berlin - Buch GmbH, Berlin
  - University Hospital Carl Gustav Carus, Dresden
  - Hautklinik Universitatsklinikum Erlangen, Erlangen
  - University Hospital Frankfurt, Frankfurt
  - SCIderm GmbH, Hamburg
  - Institute for Health Services Research in Dermatology and Nursing - IVDP, University Medical Center, Hamburg
  - Universitatsklinikum Heidelberg, Heidelberg
  - UniversitatsKlinikum Leipzig A.o.R., Leipzig
  - Comprehensive Center of Inflammatory Medicine (CCIM) University Medical Center Schleswig-Holstein, Lübeck
  - Gemeinschaftspraxis Mahlow, Mahlow
  - University Hospital Munster, Münster
  - Praxis fr Dermatologie und Venerologie, Wuppertal
- Hungary (2):
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Allergo-Derm Bakos Kft., Szolnok
- Latvia (6):
  - LTD M & M centrs, Ādaži
  - Arija's Ancane's Family Doctor Private Practice, Baldone
  - Riga 1st Hospital Skin and Sexually Transmitted Diseases Clinical Centre, Riga
  - Adoria Ltd, Riga
  - Family Doctor's Indra's Kenina's Practice, Riga
  - Health Center of Talsi Ltd, Talsi
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Radboud University Medical Centre, Nijmegen
- United Kingdom (5):
  - University Hospital of Wales, Cardiff
  - Leeds Teaching Hospitals Trust, Leeds
  - Whipps Cross University Hospital, London
  - St Helier Hospital, London
  - George Eliot Hospital, Nuneaton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Reich K, Mrowietz U, Menter A, Griffiths CEM, Bagel J, Strober B, Nunez Gomez N, Shi R, Guerette B, Lebwohl M. Effect of baseline disease severity on achievement of treatment target with apremilast: results from a pooled analysis. J Eur Acad Dermatol Venereol. 2021 Dec;35(12):2409-2414. doi: 10.1111/jdv.17520. Epub 2021 Aug 23. PMID 34255891
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690
- [Derived] Reich K, Gooderham M, Green L, Bewley A, Zhang Z, Khanskaya I, Day RM, Goncalves J, Shah K, Piguet V, Soung J. The efficacy and safety of apremilast, etanercept and placebo in patients with moderate-to-severe plaque psoriasis: 52-week results from a phase IIIb, randomized, placebo-controlled trial (LIBERATE). J Eur Acad Dermatol Venereol. 2017 Mar;31(3):507-517. doi: 10.1111/jdv.14015. Epub 2016 Dec 19. PMID 27768242

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 65 study centers in 11 countries.
Pre-assignment Details: Participants were randomized 1:1:1 to the three treatment groups. Participants were stratified according to their calculated body mass index (BMI) categories at Screening (BMI < 30 or BMI ≥ 30).
Groups:
- Placebo: Participants received placebo tablets PO BID and 2-1 ml SC saline (placebo) injections QW during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase
- Apremilast Plus Placebo Injection: Participants received apremilast 30 mg PO BID plus 2-1ml placebo SC saline injections QW during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase
- Etanercept Plus Placebo Tablet: Participants received etanercept 50 mg by SC injection QW plus placebo tablets PO BID during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase
- Placebo/Apremilast: Participants received identically matching placebo tablets by PO, BID and SC saline (placebo) injections (1mL x 2 injections SC) weekly (QW) during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase; at week 16, participants were switched to 30 mg apremilast PO BID and remained on this dose through week 104.
- Apremilast/Apremilast: Participants received apremilast 30 mg PO BID plus saline (placebo) injections (1mL x 2 injections SC) QW during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase; at week 16, participants continued on apremilast 30mg PO BID only through week 104.
- Etanercept/Apremilast: Participants received etanercept 50 mg by SC injection QW plus placebo tablets PO BID during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase; at week 16, participants discontinued etanercept and were switched to apremilast 30mg PO BID through week 104.
Period: Placebo-controlled Phase (Weeks 0-16)
Arm/Group | Placebo | Apremilast Plus Placebo Injection | Etanercept Plus Placebo Tablet | Placebo/Apremilast | Apremilast/Apremilast | Etanercept/Apremilast
Started | 84 | 83 | 83 | 0 | 0 | 0
Safety Population | 84 (Safety population includes all participants who received at least one dose of study drug.) | 83 (Safety population includes all participants who received at least one dose of study drug.) | 83 (Safety population includes all participants who received at least one dose of study drug.) | 0 | 0 | 0
Completed | 75 | 77 | 81 | 0 | 0 | 0
Not Completed | 9 | 6 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 1 | 1 | 0 | 0 | 0
Period: Apremilast Extension Phase (Weeks16-104)
Arm/Group | Placebo | Apremilast Plus Placebo Injection | Etanercept Plus Placebo Tablet | Placebo/Apremilast | Apremilast/Apremilast | Etanercept/Apremilast
Started | 0 | 0 | 0 | 73 (There are fewer participants in this period because some stopped the study at or prior to Week 16.) | 74 (There are fewer participants in this period because some stopped the study at or prior to Week 16.) | 80 (There are fewer participants in this period because some stopped the study at or prior to Week 16.)
Safety Population | 0 | 0 | 0 | 73 (Safety population includes all participants who received at least one dose of study drug.) | 74 (Safety population includes all participants who received at least one dose of study drug.) | 79 (Safety population includes all participants who received at least one dose of study drug.)
Completed | 0 | 0 | 0 | 47 | 41 | 50
Not Completed | 0 | 0 | 0 | 26 | 33 | 30
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 4 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 9 | 10 | 8
Not completed — Non-compliance With Study Drug | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 8 | 5 | 11
Not completed — Lost to Follow-up | 0 | 0 | 0 | 6 | 13 | 6
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population includes all randomized participants.
Groups:
- Apremilast Plus Placebo Injection: Participants received apremilast 30 mg PO BID plus 2-1ml SC saline (placebo) injections QW during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast Plus Placebo Injection | Etanercept Plus Placebo Tablet | Total
Number analyzed (Participants) | 84 | 83 | 83 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (14.91) | 46.0 (13.59) | 47.0 (14.07) | 45.4 (14.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 34 | 34 | 93
  Male | 59 | 49 | 49 | 157

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a 75% Improvement (Response) in the Psoriasis Area Severity Index (PASI-75) for the Comparison Between Apremilast and Placebo at Week 16 From Baseline
Description: PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy. The PASI was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The PASI score was set to missing if any severity score or degree of involvement was missing.
Time Frame: Baseline to Week 16
Population: The modified intent-to-treat (mITT) population consisted of all participants who were randomized and received at least one dose of study drug and had both a baseline PASI and at least one post-treatment PASI evaluation. Missing data imputation: Last observation carried forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Apremilast Plus Placebo Injection
Number analyzed (Participants) | 84 | 83
Percentage of participants | 11.9 | 39.8
Statistical Analysis 1: Comparison: Placebo vs Apremilast Plus Placebo Injection; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The two-sided p-value is from a CMH test stratified by the BMI at screening; Adjusted Difference = 27.5, 95% CI 2-sided [14.9 to 40.1] — The confidence interval (CI) is weighted using CMH weights according to the number of participants in the two strata

2. Secondary Outcome: Percentage of Participants Who Achieved a 75% Improvement (Response) in the Psoriasis Area and Severity Index (PASI) for the Comparison Between Etanercept 50mg SC QW and Placebo at Week 16
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: mITT population consisted of all participants who were re-randomized and received at least one dose of study drug and had both a baseline PASI and at least one post-treatment PASI evaluation. Missing data imputation: Last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Groups:
- Etanercept 50mg Plus Placebo Tablet: Participants received etanercept 50 mg by SC injection QW plus placebo tablets PO BID during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase.
Arm/Group | Placebo | Etanercept 50mg Plus Placebo Tablet
Number analyzed (Participants) | 84 | 83
percentage of participants | 11.9 | 48.2
Statistical Analysis 1: Comparison: Placebo vs Etanercept 50mg Plus Placebo Tablet; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The two-sided p-value is from a CMH test stratified by the BMI at screening; Adjusted Difference = 35.9, 95% CI 2-sided [23.3 to 48.5] — The confidence interval (CI) is weighted using CMH weights according to the number of participants in the two strata

3. Secondary Outcome: Percentage of Participants Who Achieved a Static Physician Global Assessment (sPGA) Score of Clear (0) or Almost Clear (1) With at Least 2 Points Reduction for Comparison Between Apremilast and Placebo and Etanercept and Placebo at Week 16
Description: The sPGA is an assessment by the Investigator of the overall disease severity at the time of evaluation. The sPGA is a 5-point scale ranging from 0 (clear) to 4 (severe), incorporating an assessment of the severity of the three primary signs of the disease: erythema, scaling and plaque elevation. When making the assessment of overall severity, the Investigator should factor in areas that have already been cleared (ie, have scores of 0) and not just evaluate remaining lesions for severity, ie, the severity of each sign is averaged across all areas of involvement, including cleared lesions. In the event of different severities across disease signs, the sign that is the predominant feature of the disease should be used to help determine the sPGA score.
Time Frame: Baseline and Week 16
Population: mITT population consisted of all participants who were randomized and received at least one dose of study drug and had both a baseline PASI and at least one post-treatment PASI evaluation. Missing data imputation: Last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast Plus Placebo Injection | Etanercept Plus Placebo Tablet
Number analyzed (Participants) | 84 | 83 | 83
percentage of participants | 3.6 | 21.7 | 28.9
Statistical Analysis 1: Comparison: Placebo vs Apremilast Plus Placebo Injection; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel — The p-value is from a CMH test stratified by the BMI (Body Mass Index) at screening; The p-value is from a CMH test stratified by the BMI at screening; Adjusted Difference = 18.0, 95% CI 2-sided [8.4 to 27.7] — The Confidence Interval (CI) was weighted using CMH weights according to the number of participants in the two strata
Statistical Analysis 2: Comparison: Placebo vs Etanercept Plus Placebo Tablet; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The p-value is from a CMH test stratified by the BMI (Body Mass Index) at screening; The Confidence Interval (CI) was weighted using CMH weights according to the number of participants in the two strata; Adjusted Difference = 25.2, 95% CI 2-sided [14.8 to 35.5]

4. Secondary Outcome: Percent Change From Baseline in the Affected Body Surface Area (BSA) for Comparison Between Apremilast and Placebo and Etanercept and Placebo at Week 16
Description: BSA is a measurement of involved skin. The overall BSA affected by psoriasis was estimated based on the palm area of the participant's hand (entire palmar surface or "handprint" including the fingers), which equates to approximately 1% of total body surface area. BSA percent change from baseline was determined at each visit of the study, and is calculated as 100*(post-baseline BSA - baseline BSA) / baseline BSA.
Time Frame: Baseline to Week 16
Population: mITT population consisted of all participants who were randomized and received at least one dose of study drug and had both a baseline PASI and at least one post-treatment PASI evaluation. Missing data imputation: LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Etanercept Plus Placebo Tablets: Participants received etanercept 50 mg by SC injection QW plus placebo tablets PO BID during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase
Arm/Group | Placebo | Apremilast Plus Placebo Injection | Etanercept Plus Placebo Tablets
Number analyzed (Participants) | 84 | 83 | 83
percent change | -16.3 [-23.71 to -8.81] | -47.7 [-55.20 to -40.12] | -56.1 [-63.63 to -48.59]
Statistical Analysis 1: Comparison: Placebo vs Apremilast Plus Placebo Injection; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on ANCOVA model with treatment and screening BMI category as factors and baseline value as a covariate; Difference in LS Mean = -31.40, 95% CI 2-sided [-43.33 to -19.46]
Statistical Analysis 2: Comparison: Placebo vs Etanercept Plus Placebo Tablets; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on ANCOVA model with treatment and screening BMI category as factors and baseline value as a covariate; Difference in LS Mean = -39.85, 95% CI 2-sided [-51.78 to -27.92]

5. Secondary Outcome: Percentage of Participants Who Achieved a 50% Improvement (Response) in the Psoriasis Area Severity Index (PASI-50) for Comparison Between Apremilast and Placebo and Etanercept and Placebo at Week 16
Description: PASI-50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score at Week 16. The PASI score was a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The PASI score was set to missing if any severity score or degree of involvement was missing.
Time Frame: Baseline to Week 16
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast Plus Placebo Injection | Etanercept Plus Placebo Tablet
Number analyzed (Participants) | 84 | 83 | 83
percentage of participants | 33.3 | 62.7 | 83.1
Statistical Analysis 1: Comparison: Placebo vs Apremilast Plus Placebo Injection; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — The two-sided p-value is from a CMH test stratified by the BMI at screening; Adjusted Difference = 29.4, 95% CI 2-sided [14.9 to 43.9] — The confidence interval (CI) is weighted using CMH weights according to the number of participants in the two strata
Statistical Analysis 2: Comparison: Placebo vs Etanercept Plus Placebo Tablet; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The two-sided p-value is from a CMH test stratified by the BMI at screening; Adjusted Difference = 49.8, 95% CI 2-sided [36.9 to 62.7] — The confidence interval (CI) is weighted using CMH weights according to the number of participants in the two strata

6. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score In Comparison Between Apremilast and Placebo and Etanercept and Placebo at Week 16
Description: DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the participant is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score is derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Apremilast 30mg Plus Placebo Injection: Apremilast 30 mg PO BID plus 2-1ml placebo SC saline injections QW during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase
- Etanercept 50mg Plus Placebo Tablet: Etanercept 50 mg by SC injection QW plus placebo tablets PO, BID during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase
Arm/Group | Placebo | Apremilast 30mg Plus Placebo Injection | Etanercept 50mg Plus Placebo Tablet
Number analyzed (Participants) | 81 | 79 | 80
units on a scale | -3.9 [-5.34 to -2.42] | -8.4 [-9.84 to -6.88] | -7.8 [-9.28 to -6.34]
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30mg Plus Placebo Injection; Test type: Superiority or Other; p < 0.0001, ANCOVA; Based on ANCOVA model with treatment and screening BMI category as factors and baseline value as a covariate; Difference in LS Mean = -4.48, 95% CI 2-sided [-6.82 to -2.14]
Statistical Analysis 2: Comparison: Placebo vs Etanercept 50mg Plus Placebo Tablet; Test type: Superiority or Other; p = 0.0004, ANCOVA; Based on ANCOVA model with treatment and screening BMI category as factors and baseline value as a covariate; Difference in LS Mean = -3.94, 95% CI 2-sided [-6.27 to -1.60]

7. Secondary Outcome: Change From Baseline in the Mental Component Summary (MCS) Score of the Medical Outcome Study Short Form 36-item (SF-36) Health Survey Version 2.0 in Comparison Between Apremilast and Placebo and Etanercept and Placebo at Week 16
Description: The SF-36 is a 36-item general health status instrument and consists of 8 scales: physical function (PF), role limitations-physical (RP), vitality (VT), general health perceptions (GH), bodily pain (BP), social function (SF), role limitations-emotional (RE), and mental health (MH). Scale scores range from 0 to 100, with higher scores indicating better health. Scores from the 8 scales were transformed to the norm-based scores using weights from U.S. general population to have a mean of 50 and variance = 10, with higher scores indicating better health. From these 8 scale, two overall summary scores were obtained - a Physical Component Summary score (PCS) and a Mental Component Summary score (MCS), both having the same mean of 50 and variance = 10 as noted for the individual scales for the U.S. general population, and with higher scores indicating better health. For MCS, change from baseline was calculated, where change = visit value - baseline value.
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Apremilast Plus Placebo Injection | Etanercept Plus Placebo Tablets
Number analyzed (Participants) | 81 | 80 | 80
units on a scale | 2.6 [0.72 to 4.43] | 3.5 [1.62 to 5.38] | 4.8 [2.92 to 6.67]
Statistical Analysis 1: Comparison: Placebo vs Apremilast Plus Placebo Injection; Test type: Superiority or Other; p = 0.7112, ANCOVA; Based on ANCOVA model with treatment and screening BMI category as factors and baseline value as a covariate; Difference in LS Mean = 0.93, 95% CI 2-sided [-2.05 to 3.90]
Statistical Analysis 2: Comparison: Placebo vs Etanercept Plus Placebo Tablets; Test type: Superiority or Other; p = 0.1719, ANCOVA; Based on ANCOVA model with treatment and screening BMI category as factors and baseline value as a covariate; Difference in LS Mean = 2.22, 95% CI 2-sided [-0.75 to 5.19]

8. Secondary Outcome: Percentage of Participants Who Achieved a Lattice System Physician's Global Assessment (LS-PGA) Score of Clear (0) or Almost Clear at Week 16 in Comparison Between Apremilast and Placebo and Etanercept and Placebo at Week 16
Description: The Lattice System Physician's Global Assessment is a global assessment performed by the investigator of psoriasis severity. Integrating ranges of BSA involvement with assessments of overall plaque severity (using a 4 point scale from none to marked for the signs of plaque elevation, erythema and scale), the LS-PGA produces an overall assessment of psoriasis severity on an 8-point scale, ranging from clear to very severe. To determine the final score, the lattice portion is governed by the BSA and among the plaque qualities, weights plaque elevation as most important, erythema next, and scale least.
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast Plus Placebo Injection | Etanercept Plus Placebo Tablets
Number analyzed (Participants) | 84 | 83 | 83
percentage of participants | 6.0 | 24.1 | 22.9
Statistical Analysis 1: Comparison: Placebo vs Apremilast Plus Placebo Injection; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel — The two-sided p-value is from a CMH test stratified by the BMI at screening; Adjusted Difference = 18.1, 95% CI 2-sided [7.6 to 28.6] — The confidence interval (CI) is weighted using CMH weights according to the number of participants in the two strata
Statistical Analysis 2: Comparison: Placebo vs Etanercept Plus Placebo Tablets; Test type: Superiority or Other; p = 0.0021, Cochran-Mantel-Haenszel — The two-sided p-value is from a CMH test stratified by the BMI at screening; Adjusted Difference = 16.7, 95% CI 2-sided [6.5 to 26.9] — The confidence interval (CI) is weighted using CMH weights according to the number of participants in the two strata

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During the Placebo-Controlled Phase
Description: A TEAE is an AE with a start date on or after the date of the first dose of study drug and no later than 28 days after the last dose of study drug for participants who discontinued early. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen during the study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the patient's health, including laboratory test values, regardless of etiology. Any worsening (ie, clinically significant adverse change in frequency or intensity of a preexisting condition) should be considered an AE. A serious AE (SAE) is any untoward AE that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly/birth defect, or is a condition that may jeopardize or may require intervention to prevent one of the outcomes above.
Time Frame: Week 0 to Week 16; mean duration of exposure was 14.90 weeks for placebo group, 15.13 weeks for apremilast group and 15.87 weeks for Etanercept group
Population: Safety population includes all participants who were randomized and received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Apremilast Plus Placebo Injection | Etanercept Plus Placebo Tablets
Number analyzed (Participants) | 84 | 83 | 83
participants
  Any TEAE | 45 | 59 | 44
  Any Drug-related TEAE | 17 | 27 | 21
  Any Severe TEAE | 2 | 3 | 3
  Any Serious TEAE | 0 | 3 | 2
  Any Serious Drug-related TEAE | 0 | 2 | 1
  Any TEAE Leading to Drug Interruption | 1 | 9 | 3
  Any TEAE Leading to Drug Withdrawal | 2 | 3 | 2
  Any TEAE Leading to Death | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During the Apremilast-exposure Period
Description: A TEAE in the apremilast-exposure phase is an AE with a start date on or after the date of the first dose of study drug and no later than 28 days after the last dose of study drug. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen during the study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE. A serious AE (SAE) is any untoward AE that is fatal, life-threatening, results in persistent or significant disability or incapacity, requires or prolongs existing in-patient hospitalization, is a congenital anomaly/birth defect, or is a condition that may jeopardize or may require intervention to prevent one of the outcomes listed above.
Time Frame: From the first dose of apremilast (either Week 0 for participants originally randomized to apremilast or Week 16 for those originally randomized to placebo or etanercept who were switched to apremilast at week 16) until 28 days after last apremilast dose
Population: All participants who received apremilast at any time during the study.
Measure: Number; unit: participants
Groups:
- Placebo/Apremilast: Participants received identically matching placebo tablets PO BID and SC saline (placebo) injections (1mL x 2 injections SC) QW during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase; at week 16, participants were switched to 30 mg Apremilast PO BID and remained on this dose through week 104.
- Apremilast/Apremilast: Participants received apremilast 30 mg PO BID plus saline (placebo) injections (1mL x 2 injections SC) QW during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase; at week 16, participants continued on apremilast 30mg PO BID through week 104.
- Etanercept/Apremilast: Participants received etanercept 50 mg by SC injection QW plus placebo tablets PO BID during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase; at week 16, participants were switched to apremilast 30mg PO BID through week 104.
Arm/Group | Placebo/Apremilast | Apremilast/Apremilast | Etanercept/Apremilast
Number analyzed (Participants) | 73 | 83 | 79
participants
  Any TEAE | 45 | 71 | 54
  Any Drug-related TEAE | 23 | 36 | 15
  Any Severe TEAE | 4 | 7 | 7
  Any Serious TEAE | 5 | 6 | 4
  Any Serious Drug-related TEAE | 2 | 2 | 1
  Any TEAE Leading to Drug Interruption | 8 | 13 | 7
  Any TEAE Leading to Drug Withdrawal | 3 | 7 | 2
  Any TEAE Leading to Death | 0 | 0 | 0

11. Secondary Outcome: Psoriasis Flare/Rebound
Description: Psoriasis flare is an AE and represents an atypical or unusual worsening of disease during treatment. It is defined as a sudden intensification of psoriasis requiring medical intervention or a diagnosis of new generalized erythrodermic, inflammatory, or pustular psoriasis. Rebound is an AE and is defined as a severe and sudden worsening of disease that occurs after treatment has been discontinued. This exacerbation is characterized by a PASI ≥125% of baseline or a new generalized pustular, erythrodermic, or more inflammatory psoriasis after stopping therapy.
Time Frame: Week 0 to Week 16; Placebo controlled phase
Population: Safety population includes all participants who were randomized and received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | Apremilast Plus Placebo Injection | Etanercept Plus Placebo Tablets
Number analyzed (Participants) | 84 | 83 | 83
participants
  Any psoriasis flare captured as a TEAE | 3 | 1 | 0
  Any psoriasis rebound captured as a TEAE | 0 | 0 | 0
  Those with PASI ≥125% baseline score and D/C APR | 1 | 0 | 0

12. Secondary Outcome: Psoriasis Flare/Rebound
Description: Psoriasis flare is an AE and represents an atypical or unusual worsening of disease during treatment. It is defined as a sudden intensification of psoriasis requiring medical intervention or a diagnosis of new generalized erythrodermic, inflammatory, or pustular psoriasis. Rebound is an AE and is defined as a severe and sudden worsening of disease that occurs after treatment has been discontinued. This exacerbation is characterized by a PASI ≥125% of baseline or a new generalized pustular, erythrodermic, or more inflammatory psoriasis after stopping therapy. PASI ≥125% of baseline score at any visit after the last dose date for those who discontinued within the phase.
Time Frame: From the first dose of apremilast (either Week 0 or Week 16 for participants originally randomized to placebo or etanercept who were switched at Week 16) until 28 days after the last dose of apremilast.
Population: Safety population includes all participants who were randomized and received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Placebo/Apremilast: Participants received identically matching placebo tablets by mouth (PO), twice a day (BID) and subcutaneous (SC) saline (placebo) injections (1mL x 2 injections SC) weekly (QW) during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase; at week 16, participants were switched to 30 mg Apremilast PO BID and remained on this dose through week 104.
Arm/Group | Placebo/Apremilast | Apremilast/Apremilast | Etanercept/Apremilast
Number analyzed (Participants) | 73 | 83 | 79
participants
  Any psoriasis flare captured as a TEAE | 1 | 4 | 0
  Any psoriasis rebound captured as a TEAE | 1 | 2 | 7
  Those with PASI ≥125% baseline score and D/C APR | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the 16-week placebo-controlled period and up to week 104 during the apremilast exposure period for all participants who were randomized or switched to apremilast at any time during the course of the study.
Description: The mean duration of exposure was 14.90 weeks, 15.13 weeks, and 15.87 weeks for participants randomized to the placebo, apremilast 30 BID, and etanercept 50 mg every week treatment groups, respectively during the placebo controlled phase. The mean duration of exposure to apremilast 30 mg BID during the apremilast exposure period was 69.13 weeks.
Groups:
- Placebo (Week 0-16): Participants received placebo tablets PO BID and 2-1 milliliter (ml) SC saline (placebo) injections QW during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase
- Apremilast Plus Placebo Injection (Week 0-16): Participants received Apremilast 30 mg PO BID plus 2-1ml SC saline (placebo) injections QW during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase
- Etanercept Plus Placebo Tablets (Week 0-16): Participants received etanercept 50 mg by SC injection QW plus placebo tablets PO BID during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase
- Placebo/APR 30mg (Apremilast Exposure Phase) Weeks 16-104: Participants received identically matching placebo tablets by mouth (PO), twice a day (BID) and subcutaneous (SC) saline (placebo) injections (1mL x 2 injections SC) weekly (QW) during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase; at week 16, participants were switched to 30 mg Apremilast PO BID and remained on this dose through week 104.
- APR/APR 30 mg (Apremilast Exposure Phase) Weeks 0-104: Participants received apremilast 30 mg PO BID plus saline (placebo) injections (1mL x 2 injections SC) QW during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase; at week 16, participants continued on apremilast 30mg PO BID through week 104.
- Etanercept/APR 30mg (Apremilast Exposure Phase) Weeks 16-104: Participants received etanercept 50 mg by SC injection QW plus placebo tablets PO BID during the 16-week randomized, double-blind, double-dummy, placebo-controlled phase; at week 16, participants were switched to apremilast 30mg PO BID through week 104.
Arm/Group | Placebo (Week 0-16) | Apremilast Plus Placebo Injection (Week 0-16) | Etanercept Plus Placebo Tablets (Week 0-16) | Placebo/APR 30mg (Apremilast Exposure Phase) Weeks 16-104 | APR/APR 30 mg (Apremilast Exposure Phase) Weeks 0-104 | Etanercept/APR 30mg (Apremilast Exposure Phase) Weeks 16-104
Serious Adverse Events (participants affected / at risk) | 0/84 | 3/83 | 2/83 | 5/73 | 6/83 | 4/79
Other Adverse Events (participants affected / at risk) | 25/84 | 41/83 | 27/83 | 30/73 | 52/83 | 32/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0-16) (N=84) | Apremilast Plus Placebo Injection (Week 0-16) (N=83) | Etanercept Plus Placebo Tablets (Week 0-16) (N=83) | Placebo/APR 30mg (Apremilast Exposure Phase) Weeks 16-104 (N=73) | APR/APR 30 mg (Apremilast Exposure Phase) Weeks 0-104 (N=83) | Etanercept/APR 30mg (Apremilast Exposure Phase) Weeks 16-104 (N=79)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Anogenital warts (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Pneumocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0-16) (N=84) | Apremilast Plus Placebo Injection (Week 0-16) (N=83) | Etanercept Plus Placebo Tablets (Week 0-16) (N=83) | Placebo/APR 30mg (Apremilast Exposure Phase) Weeks 16-104 (N=73) | APR/APR 30 mg (Apremilast Exposure Phase) Weeks 0-104 (N=83) | Etanercept/APR 30mg (Apremilast Exposure Phase) Weeks 16-104 (N=79)
Nausea (Gastrointestinal disorders) | 1 | 9 | 4 | 5 | 12 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 9 | 1 | 13 | 12 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 6 | 2 | 5 | 9 | 1
Nasopharyngitis (Infections and infestations) | 8 | 4 | 8 | 4 | 5 | 5
Headache (Nervous system disorders) | 3 | 11 | 5 | 5 | 12 | 3
Tension Headache (Nervous system disorders) | 4 | 5 | 3 | 3 | 5 | 1
Toothache (Gastrointestinal disorders) | 1 | 4 | 2 | 2 | 5 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 2 | 3 | 6 | 2
Rhinitis (Infections and infestations) | 1 | 4 | 4 | 1 | 6 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 3 | 0 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 4 | 6 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 4 | 4
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 3 | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4 | 1 | 6 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 1 | 5 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 2 | 5 | 0
Rebound psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 7
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 12 months since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.